CLINICAL TRIAL: NCT02573077
Title: A Prospective, Observational Study Measuring Sodium Improvement and Outcomes in Cancer Patients Treated for Moderate to Severe Hyponatremia Secondary to SIADH in Italy
Brief Title: An Observational Study Measuring Outcomes in Cancer Patients Treated for Moderate to Severe Hyponatremia in Italy
Acronym: ASSERT
Status: Completed | Type: Observational
Sponsor: Otsuka Pharmaceutical Europe Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: OPEL/2014/067
Record Dates: First submitted 2015-10-06; First posted 2015-10-09 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Hyponatremia; Syndrome of Inappropriate ADH (SIADH) Secretion; Cancer
Keywords: Hyponatremia due to SIADH; Cancer
MeSH Terms: conditions — Hyponatremia; Inappropriate ADH Syndrome; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This observational, prospective, non-interventional study will include cancer patients who need a treatment for hyponatraemia secondary to SIADH. Patients will be prescribed treatment(s) according with the clinical practice regardless of the patient participation in the study. The purpose of this NIS is to collect additional scientific and clinical information that can help in describing the characteristics of cancer patients with hyponatraemia secondary to SIADH, the current management of hyponatremia, the therapies to keep under control serum [Na+] and the guidelines for the management of this population in Italy.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years;
2. Male or female patients with a cytologically or histologically documented cancer diagnosis;
3. Moderate to severe hyponatremia: Na+ level cut off: [Na+] < 130 mmol/L;
4. Physician diagnosed Moderate to severe hyponatremia secondary to SIADH (clinical or laboratory determined as per normal routine practice of treating physician);
5. No use of diuretic agents within the week prior to evaluation;
6. Willingness to participate in the study; subjects must give their written consent to participate.

Exclusion Criteria:

1. Use of concomitant medications including demeclocycline and/or urea, by themselves or in combination with fluid restriction;
2. Subject is currently participating in a clinical trial in which the investigational medicinal product aims to treat the causes or symptoms of hyponatremia;
3. Life expectancy is lower than 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This non-interventional study will include cancer patients who need a treatment for hyponatremia secondary to SIADH in one of the hospitals participating in the study.
Sampling Method: Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-12-13 (Actual); Study Completion 2017-12-13 (Actual)

PRIMARY OUTCOMES:
Change in serum [Na+] | 1 month and 6 months
  Change in serum [Na+] from the baseline visit to the end of the first month or sixth month of the observational period or until earlier discontinuation from the study

SECONDARY OUTCOMES:
EQ-5D to measure quality of life | From baseline up to 6 months
  Will be assessed at baseline and at subsequent visits (falling within routine clinical practice) until 6 months.
  EQ-5D EQ-5D is a standardised measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal.
EORTC QLQ-C30 to measure quality of life | From baseline up to 6 months
  Will be assessed at baseline and at subsequent visits (falling within routine clinical practice) until 6 months.
  EORTC QLC-C30: European Organisation for Research and Treatment of Cancer (EORTC) Study Group on Quality of Life has developed the EORTC QLQ-C30 questionnaire consisting in a modular system for assessing the quality of life of cancer patients in clinical research.
ECOG PS to assess progress of the disease | From baseline up to 6 months
  Will be assessed at baseline and at subsequent visits (falling within routine clinical practice) until 6 months.
  The Eastern Cooperative Oncology Group (ECOG) performance status is a scale used to assess how a patient's disease is progressing, assess how the disease affects the daily living abilities of the patient, and determine appropriate (oncology) treatment and prognosis.
Measure of cognitive impairment: mini-mental state examination (MMSE) | From baseline up to 6 months
  Will be assessed at baseline and at subsequent visits (falling within routine clinical practice) until 6 months.
  The mini-mental state examination (MMSE) or Folstein test is a sensitive, valid and reliable 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment.
Time to chemotherapy (days) | Longitudinal (up to 6 months)
Length of stay (days) | Longitudinal (up to 6 months)
Readmission (number of readmissions) | Longitudinal (up to 6 months)
  will be used to evaluate rate of readmissions among this population
Survival status (%) | 6 months
  Will be used to evaluate overall survival (%) among this population after 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Department, Study Director — Otsuka Europe
Locations (20):
- Italy (20):
  - Ancona
  - Aosta
  - Bari
  - Cagliari
  - Cosenza
  - Florence
  - Genova
  - Messina
  - Milan
  - Napoli
  - Negrar
  - Novara
  - Palermo
  - Parma
  - Perugia
  - Piacenza
  - Pisa
  - Roma
  - Varese
  - Verona